CLINICAL TRIAL: NCT06352437
Title: Safety, Tolerability and Pharmacokinetics of Single Subcutaneous Doses of BI 3034701 in Healthy Male Volunteers (Part A) and of Multiple Rising Subcutaneous Doses in Otherwise Healthy Male and Female Volunteers With Obesity/Overweight (Part B)
Brief Title: A Study to Test How Well Different Doses of BI 3034701 Are Tolerated by Healthy Men and People With Overweight or Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1507-0001; 2023-508767-79-00 (Registry Identifier: CTIS); U1111-1302-5933 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2024-04-03; First posted 2024-04-08 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- Part A: BI 3034701 dose group 1 (Experimental)
- Part A: BI 3034701 dose group 2 (Experimental)
  Interventions: Drug: BI 3034701
- Part A: BI 3034701 dose group 3 (Experimental)
  Interventions: Drug: BI 3034701
- Part A: BI 3034701 dose group 4 (Experimental)
  Interventions: Drug: BI 3034701
- Part A: BI 3034701 dose group 5 (Experimental)
  Interventions: Drug: BI 3034701
- Part A: BI 3034701 dose group 6 (Experimental)
  Interventions: Drug: BI 3034701
- Part A: BI 3034701 dose group 7 (Experimental)
- Part A: BI 3034701 dose group (Experimental)
  Interventions: Drug: BI 3034701
- Part A: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo matching BI 3034701
- Part B: BI 3034701 dose group 1 (Experimental)
  Interventions: Drug: BI 3034701
- Part B: BI 3034701 dose group 2 (Experimental)
  Interventions: Drug: BI 3034701
- Part B: BI 3034701 dose group 3 (Experimental)
  Interventions: Drug: BI 3034701
- Part B: BI 3034701 dose group 4 (Experimental)
  Interventions: Drug: BI 3034701
- Part B: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo matching BI 3034701

INTERVENTIONS:
Drug: BI 3034701 — BI 3034701
  Arms: Part A: BI 3034701 dose group; Part A: BI 3034701 dose group 2; Part A: BI 3034701 dose group 3; Part A: BI 3034701 dose group 4; Part A: BI 3034701 dose group 5; Part A: BI 3034701 dose group 6; Part B: BI 3034701 dose group 1; Part B: BI 3034701 dose group 2; Part B: BI 3034701 dose group 3; Part B: BI 3034701 dose group 4
Drug: Placebo matching BI 3034701 — Placebo matching BI 3034701
  Arms: Part A: Placebo; Part B: Placebo

SUMMARY:
This study is open to healthy people and people with overweight or obesity. It has 2 parts. Part A is open to healthy men between 18 and 55 years of age. Part B is open to people between 18 and 65 years of age with overweight or obesity who are otherwise healthy.

The purpose of this study is to find out how well different doses of BI 3034701 are tolerated by healthy men (Part A) and people with overweight or obesity (Part B). Another goal of this study is to find out how different doses of BI 3034701 are taken up in the blood.

Participants get different doses of BI 3034701 or placebo as an injection under the skin. In Part A, every participant gets a single dose. In Part B, every participant gets several doses of BI 3034701 or placebo. In this study, BI 3034701 is given to humans for the first time.

Participants in Part A are in the study up to 10 weeks. During this time, they visit the study site 8 times. Participants in Part B are in the study for about 5 months. They visit the study regularly. At some of the visits, participants in both parts stay at the study site for up to 5 nights. During the study, the doctors collect information on any health problems of the participants.

ELIGIBILITY:
Inclusion Criteria:

1. Part A: healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests.

   Part B: healthy male or female subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests.
2. Part A: age of 18 to 55 years (inclusive). Part B: age 18 to 65 years (inclusive).
3. Parts A and B: Signed and dated written informed consent in accordance with the International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use - Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial.
4. Further inclusion criteria apply

Exclusion Criteria:

1. Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator.
2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm).
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance and, in particular:

   * Alanine aminotransferase (ALT) above upper limit of normal (ULN) + 20%
   * Aspartate aminotransferase (AST) above ULN + 20%
   * Gamma-Glutamyl-Transferase (GGT) above ULN + 20%
   * Lipase or amylase above ULN + 20%
   * Bilirubin above 1.2x ULN (except for cases of Gilbert's Syndrome)
   * Estimated glomerular filtration rate (eGFR) < 80 mL/min/1.73 m²
4. Any evidence of a concomitant disease assessed as clinically relevant by the investigator.
5. Further exclusion criteria apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2025-10-07 (Actual); Study Completion 2025-10-07 (Actual)

PRIMARY OUTCOMES:
Part A and Part B: Occurrence of any treatment-emergent adverse event assessed as drug-related by the investigator | up to 48 days for Part A and up to 130 days for Part B.

SECONDARY OUTCOMES:
Part A: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) following a single dose of BI 3034701 | up to 48 days.
Part A: Maximum measured concentration of the analyte in plasma (Cmax) following a single dose of BI 3034701 | up to 48 days.
Part B: Area under the concentration-time curve in plasma over the dosing interval of 0 to 168 hours (AUCtau) following multiple doses of BI 3034701 | up to 130 days.
Part B: Maximum measured concentration of the analyte in plasma (Cmax) following multiple doses of BI 3034701 | up to 130 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Research Organisation GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com